CLINICAL TRIAL: NCT00950222
Title: Impact of Imipenem With Amikacin Pharmacokinetic and Pharmacodynamic
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P061014; CRC06049 (Other: CRC)
Record Dates: First submitted 2009-07-28; First posted 2009-07-31 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Intensive care unit; Ventilator associated pneumonia; Gram negative bacilli infection; Empirical antibiotic therapy; Pharmacokinetic / pharmacodynamic; Imipenem; Amikacin; Gram negative bacilli
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Gram-Negative Bacterial Infections | interventions — Imipenem; Amikacin; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1:Imipenem/Amikacin (Experimental): patients will receive as empirical therapy for VAP imipenem associated with amikacin.After primary outcome measure, antibiotic therapy will be left at the discretion of the physician in charge of the patient.
  Imipenem: recommended usual dosage for VAP treatment, IV (in the vein), every 8 hours
  Amikacin: recommended usual dosage for VAP treatment (20mg/kg), IV (in the vein), single dose (at H0) for the 48 first hours of treatment
  Interventions: Drug: Imipenem/Amikacin

INTERVENTIONS:
Drug: Imipenem/Amikacin — patients will received as empirical therapy for VAP imipenem associated with amikacin.
  Other Names: Therapy for VAP imipenem associated with amikacin

SUMMARY:
The study is a prospective open trial conducted in 4 centers, and designed to determine if pharmacokinetic (PK) and pharmacodynamic (PD) parameters of imipenem, associated with amikacin as empirical therapy, impact microbiological and clinical outcome of patients with Gram negative bacilli (GNB) ventilator-associated pneumonia (VAP).

DETAILED DESCRIPTION:
Inappropriate initial antibiotherapy increases mortality of many serious infections. This is the case for ventilator-associated pneumonia, frequently occurring during intensive care unit (ICU) hospitalization, and whose 48 first hours of treatment are decisive.

It is well established that pharmacokinetic and pharmacodynamic parameters of antibiotics are correlated with their clinical and microbiological effectiveness. However in ICU patients, pharmacokinetic parameters of antibiotics suffer great variations, and bacteria responsible for these infections are usually less sensitive to antibiotics, especially Gram negative bacilli (GNB). An important pharmacodynamic variability may occur at the initial phase of the antibiotic treatment, decisive for the infection's outcome.

We propose to evaluate the correlation between pharmacokinetic and pharmacodynamic profile of the empirical antibiotic therapy and the microbiological and clinical outcome of VAP.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Mechanical ventilation for more than 48 hours
3. Clinical suspicion of VAP defined by a new persistent radiological infiltrate and one of the following signs: purulent tracheal aspirations, or temperature of 38°3 or higher, or leucocyte count > 10000/ml
4. Risk of multi resistant bacteria defined as follows: at least 6 days of mechanical ventilation or antibiotic treatment in the 15 previous days
5. Distal pulmonary secretion sample obtained beforehand for microbiological diagnosis by bronchoalveolar lavage via bronchoscopy or blinded protected telescoping catheter via bronchoscopy or blindly
6. Presence of GNB on direct examination of the distal pulmonary secretion sample
7. Realization of a preliminary medical examination. 8- Written inform consent from the patient or relatives. The consent may be obtained after the enrollment if the patient is not able to give consent and if there is no relatives

Exclusion Criteria:

1. Time between distal pulmonary secretion sample taking and the 1st administration of imipenem exceeding 24 hours
2. Pregnancy
3. Severely impaired renal function (creatinine clearance lower than 10 mL/mn or renal replacement therapy)
4. Allergy to imipenem or amikacin
5. Treatment in progress with imipenem or amikacin
6. Death expected within 48 hours following diagnosis of VAP
7. Myasthenia
8. Simultaneous administration of others aminoglycosides
9. Association with intravenous polymyxin or botulinum toxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Variation of numeration (cfu per ml) of GNB, for whom culture of pulmonary samples are positive (higher than defined thresholds), between the quantitative endotracheal aspiration (QAE) obtained at H0 (initiation of treatment) and QAE obtained at H48 | Hour 48

SECONDARY OUTCOMES:
To describe imipenem and amikacin PK parameters as empirical therapy in ICU patients treated for VAP | Hour 24
To describe imipenem and amikacin PD parameters as empirical therapy in ICU patients treated for VAP | Hour 24
To determine the proportion of patients for whom the pharmacodynamic targets suggested in the literature for aminoglycosides and beta lactams are achieved | Hour 24
To identify sources of variability of imipenem and amikacin PK/PD parameters in ICU patients with VAP | Hour 24
To assess the impact of imipenem and amikacin PK/PD parameters on GNB eradication at day 3 | Day 3
To assess the impact of imipenem and amikacin PK/PD parameters variability on the CPIS, clinical score of VAP, measured 48 hours after initiation of the treatment | Hour 48
To assess the impact of imipenem and amikacin PK/PD parameters on the time necessary to observe a CPIS lower or equal to 6 | Day 8
To assess the impact of imipenem and amikacin PK/PD parameters on clinical evolution of the VAP after 7 days of antibiotic treatment | Day 8
To assess the impact of imipenem and amikacin PK/PD parameters on serum procalcitonin levels evolution between the initiation of the treatment and 48 hours after the initiation of the treatment of the VAP | Hour 48
To assess the impact of imipenem and amikacin PK/PD parameters on mortality at day 28 (Day 28) 11- to assess the impact of imipenem and amikacin PK/PD parameters on VAP relapse | Day 28
To study emergence of less sensitive bacteria to imipenem and/or amikacin, 48 hours after the initiation of the antibiotic treatment, among GNB isolated in endotracheal aspiration before initiation of this treatment | Hour 48
To study emergence in the tracheal and digestive flora of micro-organisms resistant to imipenem after the first 48 hours of treatment by imipenem | Hour 48

CONTACTS AND LOCATIONS:
Overall Officials: Olivier PAJOT, MD, Principal Investigator — HOPITAL ARGENTEUIL
Locations (1):
- Victor Dupouy Hospital, Argenteuil, France

REFERENCES:
- [Derived] Burdet C, Pajot O, Couffignal C, Armand-Lefevre L, Foucrier A, Laouenan C, Wolff M, Massias L, Mentre F. Population pharmacokinetics of single-dose amikacin in critically ill patients with suspected ventilator-associated pneumonia. Eur J Clin Pharmacol. 2015 Jan;71(1):75-83. doi: 10.1007/s00228-014-1766-y. Epub 2014 Oct 21. PMID 25327505
- [Derived] Couffignal C, Pajot O, Laouenan C, Burdet C, Foucrier A, Wolff M, Armand-Lefevre L, Mentre F, Massias L. Population pharmacokinetics of imipenem in critically ill patients with suspected ventilator-associated pneumonia and evaluation of dosage regimens. Br J Clin Pharmacol. 2014 Nov;78(5):1022-34. doi: 10.1111/bcp.12435. PMID 24903189